CLINICAL TRIAL: NCT04946682
Title: Optimal Encephalitis/Meningitis Roadmap Via Precise Diagnosis and Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wen-hong Zhang (Other)
Responsible Party: Sponsor-Investigator, Wen-hong Zhang, chairman of the infectious disease department, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IMPROVE
Record Dates: First submitted 2021-05-27; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Encephalitis; Meningitis; Meningoencephalitis; Next-Generation Sequencing; Polymerase Chain Reaction
MeSH Terms: conditions — Encephalitis; Meningitis; Meningoencephalitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of mNGS (Experimental)
  Interventions: Diagnostic Test: Types of etiological diagnostic methods
- Group of PCR (Experimental)
  Interventions: Diagnostic Test: Types of etiological diagnostic methods

INTERVENTIONS:
Diagnostic Test: Types of etiological diagnostic methods — In Group of mNGS, all patients will be tested by meta next generation sequncing on admission, while patients in Group of PCR will be tested by polymerase chain reaction in accordance with the method in the guidelines.

SUMMARY:
Encephalitis and meningitis are serious central nervous system diseases. There is currently a lack of comprehensive and accurate diagnosis and treatment pathways. Therefore, we conducted this multicenter, prospective, and randomized controlled study. It was designed to evaluate the diagnostic performance and its impact on the outcomes of the patients enrolled. As such, we came to the results of the optimal process of diagnosis and treatment strategy of encephalitis/meningeal syndromes with improved effective treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected meningitis : the patient has a new fever (>38.5℃), accompanied by ≥1 of the following manifestations：

  1. Stiff neck
  2. Change in state of consciousness
  3. Other signs of meningitis: such as meningeal irritation.
* Patients with suspected encephalitis: Unexplained changes in the state of consciousness for more than 24 hours (including lethargy, agitation, personality changes, etc.) or accompanied by recent memory impairment, with the following ≥1 manifestations:

  1. Fever during the course of the disease (≥ 38℃); (oral temperature)
  2. Convulsions or focal neurological symptoms;
  3. Increase in the number of cerebrospinal fluid cells (>4*10^6/L);
  4. Abnormal EEG that meets the manifestations of encephalitis and cannot be attributed to other reasons
  5. Imaging suggests encephalitis (CT or MRI)
* Have not received effective anti-infective treatment yet
* Have an identifiable address and live in the area during treatment.
* Suspected encephalitis/meningitis patients who are willing to participate in trial treatment and follow-up and can give informed consent (if the subject is illiterate, sign or hearing consent is required).
* Willing to comply with follow-up research procedures.

Exclusion Criteria:

* Known breastfeeding or pregnancy
* Failure to comply with treatment or follow-up time;
* The researcher believes that there are any conditions (social or medical) that allow subjects to participate in unsafe;
* Participating in other clinical studies
* Insufficient cerebrospinal fluid or blood samples
* Clinically diagnosed infections, tumors or other neurological diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-04-14 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
The change Modified Rankin Scale (mRS) at 1 year | mRS should be measured at 1 year
  The Modified Rankin Scale at 1 year Grade Description 0 No symptoms
  1. Minor symptoms not interfering with lifestyle
  2. Symptoms that lead to some restriction in lifestyle, but do not interfere with the patients' ability to look after themselves
  3. Symptoms that restrict lifestyle and prevent totally independent living
  4. Symptoms that clearly prevent independent living, although the patient does not need constant care and attention
  5. Totally dependent, requiring constant help day and night

SECONDARY OUTCOMES:
Mortality rate at 1 year | Mortality rate at 1 year
  Mortality rate at 1 year

OTHER OUTCOMES:
Time required from 1 day of admission to the initiation of the target treatment | Baseline (The time point of getting the target treatment - the time point of admission)
  The time required for the patients to get the target treatment from 1 day of admission.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Nanjing Hospital of Chinese Medicine Affiliated to Nanjing University of Chinese Medicine, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi No.5 People's Hospital, Wuxi, Jiangsu
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Blue Cross Brain Hospital, Shanghai, Shanghai Municipality
  - People's Hospital of Zhuji, Zhejiang Province, Zhuji, Zhejiang

REFERENCES:
- [Derived] Zhang Y, Zhang H, Deng B, Lin K, Jin L, Liu X, Zhang Y, Chen X, Zhang Y, Lu S, Huang H, Wang Q, Feng T, Zhao W, Xue Q, Chen R, Zhang J, Qian X, Chen L, Ai J, Chen X, Zhang W. Optimal encephalitis/meningitis roadmap via precise diagnosis and treatment (IMPROVE): a study protocol for a randomized controlled trial. BMC Infect Dis. 2022 Jan 8;22(1):40. doi: 10.1186/s12879-021-06943-6. PMID 34998377